CLINICAL TRIAL: NCT00783952
Title: Validation of Mixed Venous Blood Oxygen Saturation Obtained With a Novel Mathematical Equation Using Arterial Oxygen Saturation and Various Local Tissue Oxygen Saturations.
Brief Title: Validation of Mixed Venous Blood Oxygen Saturation Obtained With a Novel Mathematical Equation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit subjects
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert M. Kacmarek, Professor of Anesthesia, Director of Respiratory Care Services, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2008-P-000420
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Mixed Venous Oxygen Saturation; Tissue Oxygenation
Keywords: Mixed venous oxygen saturation; Tissue oxygenation; Near infrared spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Mixed venous oxygen saturation measurement obtained from blood drawn from a pulmonary artery catheter.Calculation of mixed venous oxygen saturation from the measurement of peripheral oxygen saturations using multiple Cerebral/Somatic Tissue Oximeter device probes
  Interventions: Device: Cerebral/Somatic Tissue Oximeter device; Device: Pulmonary artery catheter

INTERVENTIONS:
Device: Cerebral/Somatic Tissue Oximeter device — Measurement of tissue oxygen saturation and simultaneous sampling for blood gas analysis.
  Four sensors of the 'Cerebral/Somatic Tissue Oximeter' device will be placed on subject's both sides of the forehead, palm and calf area. Simultaneously, blood samples will be drawn from the pulmonary artery catheter and arterial line for blood gas analyses. The values obtained from the device measurements will be used in a new equation to calculate the mixed venous oxygen saturation. The calculated value will be compared to the real value from the blood gas analysis for accuracy.
Device: Pulmonary artery catheter — Blood will be drawn form the pulmonary artery catheter for measurement of mixed venous oxygen saturation.

SUMMARY:
The purpose of this study is to test a new way to measure the oxygen level in the mixed venous blood system (the system that carries blood collected from all over the body to the heart), which is a very important monitoring tool for the overall oxygen delivery to all our tissues. This new way measures the oxygen level in the mixed venous blood from outside the body, instead of measuring from the inside through a catheter (a thin, flexible plastic tube) that is placed by breaking the skin.

DETAILED DESCRIPTION:
Study terminated because of inability to recruit subjects

ELIGIBILITY:
Inclusion Criteria:

* Patients already being monitored by a pulmonary artery catheter and an arterial line

Exclusion Criteria:

* Patients with severe heart failure
* Patients with carbon monoxide or thiocyanate poisoning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kacmarek, PhD, RRT, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mixed Venous Oxygen and Calculation of Saturation: Blood will be drawn form the pulmonary artery catheter for measurement of mixed venous oxygen saturation.Measurement of tissue oxygen saturation and simultaneous sampling for blood gas analysis.
  Four sensors of the 'Cerebral/Somatic Tissue Oximeter' device will be placed on subject's both sides of the forehead, palm and calf area. Simultaneously, blood samples will be drawn from the pulmonary artery catheter and arterial line for blood gas analyses. The values obtained from the device measurements will be used in a new equation to calculate the mixed venous oxygen saturation. The calculated value will be compared to the real value from the blood gas analysis for accuracy.
Period: Overall Study
Arm/Group | Mixed Venous Oxygen and Calculation of Saturation
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Pulmonary Artery Catheters and Arterial Lines: Patients with pulmonary artery catheters and arterial lines
  'Cerebral/Somatic Tissue Oximeter' device: Measurement of tissue oxygen saturation and simultaneous sampling for blood gas analysis.
  Four sensors of the 'Cerebral/Somatic Tissue Oximeter' device will be placed on subject's both sides of the forehead, palm and calf area. Simultaneously, blood samples will be drawn from the pulmonary artery catheter and arterial line for blood gas analyses. The values obtained from the device measurements will be used in a new equation to calculate the mixed venous oxygen saturation. The calculated value will be compared to the real value from the blood gas analysis for accuracy.
Arm/Group | Patients With Pulmonary Artery Catheters and Arterial Lines
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Determining the Accuracy of Mixed Venous Oxygen Saturation Obtained With a Novel Mathematical Equation Using Arterial Oxygen Saturations and Various Local Tissue Oxygen Saturations.
Description: Four sensors of the 'Cerebral/Somatic Tissue Oximeter' device will be placed on subject's both sides of the forehead, palm and calf area. Simultaneously, blood samples will be drawn from the pulmonary artery catheter and arterial line for blood gas analyses. The values obtained from the device measurements will be used in a new equation to calculate the mixed venous oxygen saturation. The calculated value will be compared to the real value from the blood gas analysis for accuracy.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Groups:
- Patients With Cerebral/Somatic Tissue Oximeter Device: Measurement of tissue oxygen saturation and simultaneous sampling for blood gas analysis.
  Four sensors of the 'Cerebral/Somatic Tissue Oximeter' device will be placed on subject's both sides of the forehead, palm and calf area. Simultaneously, blood samples will be drawn from the pulmonary artery catheter and arterial line for blood gas analyses. The values obtained from the device measurements will be used in a new equation to calculate the mixed venous oxygen saturation. The calculated value will be compared to the real value from the blood gas analysis for accuracy.
Arm/Group | Patients With Pulmonary Artery Catheters and Arterial Lines | Patients With Cerebral/Somatic Tissue Oximeter Device
Number analyzed (Participants) | 8 | 8
percentage of oxygen saturation | 47.6 (8.0) | 61.0 (8.2)

ADVERSE EVENTS:
Arm/Group | Patients With Pulmonary Artery Catheters and Arterial Lines
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes